CLINICAL TRIAL: NCT00042510
Title: Open-Label,Multicenter Study of G17DT Immunogen in Combination w/ Cisplatin and 5-FU in Subjects w/ Metastatic or Locally Recurrent Gastric or Gastroesophageal Cancer Previously Untreated With Chemotherapy.
Brief Title: Safety and Efficacy of G17DT Immunogen in the Treatment of Gastric and Gastroesophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Advances Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC4
Record Dates: First submitted 2002-07-31; First posted 2002-08-01 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Stomach Neoplasms; Esophageal Neoplasms
Keywords: Gastroesophageal cancer; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Group (Experimental): 500µg G17DT administered on Weeks 1, 5 and 9 and an additional treatment at Week 25. Cisplatin was administered every 4 weeks on the first day of each treatment cycle as a 1 to 3 hour intravenous infusion at a dose of 100mg/m^2. 5-FU was administered every 4 weeks during the first 5 days of each cycle as a continuous intravenous infusion at a dose of 1,000 mg/m^2/d.
  Interventions: Biological: Treatment group

INTERVENTIONS:
Biological: Treatment group

SUMMARY:
This study will test whether the G17DT Immunogen, when administered in combination with chemotherapy, is an effective and safe treatment for gastric cancer.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis with gastric or gastroesophageal cancer
* Karnofsky performance status score of at least 70
* Life expectancy of at least 3 months

Exclusion criteria:

* Prior treatment with chemotherapy or anticancer immunotherapy
* Bone marrow transplant within past year
* Chronic use of corticosteroids, except for inhaled corticosteroids used for asthma or chronic obstructive pulmonary disease
* Central nervous system metastases
* Immunodeficiency
* Hypercalcemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2000-08; Primary Completion 2003-02 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of G17DT in combination with cisplatin and 5-FU chemotherapy on tumor response assessed by radiographic means. | Through Week 29

SECONDARY OUTCOMES:
To evaluate the clinical efficacy of G17DT in combination with cisplatin and 5-FU chemotherapy as measured by time to disease progression, best overall response and survival. | Through Week 29

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer A Ajani, M.D., Principal Investigator — U.S. studies; Vladimir Moiseyenko, M.D., Ph.D, Principal Investigator — Non U.S. studies